CLINICAL TRIAL: NCT02030314
Title: The Management of Resistant Hypertension in Kidney Transplant Patients Using Chlorthalidone
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The patient population changed. Unable to find patients that meet study criteria
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20002960
Record Dates: First submitted 2013-12-19; First posted 2014-01-08 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Resistant Hypertension in Kidney Transplant Patients
Keywords: Chlorthalidone; Resistant Hypertension; Kidney Transplant Patients
MeSH Terms: interventions — Chlorthalidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chlorthalidone, resistant high blood pressure (Experimental): if Furosemide dose is 40 mg per day, start Chlorthalidone 12.5 mg per day if Furosemide dose is 80 mg per day, start Chlorthalidone 25 mg per day
  Interventions: Drug: Chlorthalidone

INTERVENTIONS:
Drug: Chlorthalidone — treatment of resistant hypertension in kidney transplant patients
  Other Names: Thalitone

SUMMARY:
Chlorthalidone might offer an effective, safe and inexpensive anti-hypertensive treatment for kidney transplant patients who have resistant hypertension on multi-drug therapy. We will collect initial data on the safety and efficacy of Chlorthalidone in the treatment of patients with resistant hypertension.

To Examine the efficacy of chlorthalidone as an anti-hypertensive agent in the treatment of resistant hypertension among stable kidney transplant recipients

DETAILED DESCRIPTION:
The study involves transplant recipients presenting to the transplant Clinic Gateway 7th floor with resistant hypertension. The initial contact will take place in the transplant clinic study consist of approximately eight out patient visits over a 8 week period: Screening, and follow-up visits will be conducted at the Clinical Research Services (CRS) Unit. The Baseline (Week 1), Visit 1 Enrollment (Week 1) Day 1 and 2, Visit 2, (Week 3) Day 1 and 2, and Visit 3 End of Study, (Week 7) Day 1 and 2. Additional visits maybe required to accommodate adverse reactions. The study will require approximately four (4) time points where blood pressure, pulse and weight is obtained, safety blood collections approximately 2-3 tablespoons drawn by venipuncture and 24 hour urine collection periods. Home blood pressure readings will be required at two (2) time points during the study. The subject will be required to stop taking current medications for seven weeks, take study medication for 6 weeks and report adverse reactions and concomitant medications at each visit.

During the Enrollment visit, the subject will be identified, informed consent obtained, demographic characteristics, past medical history, co-morbid illnesses, current medications, and home and office blood pressures will be recorded to assess for eligibility criteria. This data will be collected prospectively by the investigators.

Initial clinical assessment at the time of the patient's screening visit will be performed at the outpatient testing center in the transplant clinic. A three day window will be allowed for all visits. The following measurements will occur at this visit: Biometric measurements: vitals ( blood pressure and pulse) body weight, EKG, Arm circumference, confirmation of hypertension by 24-h ABPM , urine studies: 24 hour urine collection and evaluation, safety, 8-10AM sitting upright Plasma Aldosterone/Renin Ratio, clinical safety laboratory test: bone morphogenetic protein, Mg/phosphorus level, Parathyroid hormone, vitamin D level and HbA1c, review and document concomitant medications, including current furosemide prescription. Subjects who meet the inclusion criteria and none of the exclusion criteria will start Baseline (Week 1) Measurements.

At Baseline (Week 1) the current furosemide prescription will be documented and discontinued. This will begin the washout period. The washout period will continue for one week. At the end of the washout period the subject will be instructions to return to the CRS unit for Visit 1 Enrollment measurements.

Visit 1 Enrollment Measurements Week 1, Day 1, include the following measurements: Biometric measurements: Body Weight, confirmation of hypertension by 24-h ABPM Urine studies: start 24 hour Urine collection, safety laboratory evaluations: bone morphogenetic protein , document concomitant medications, and adverse reactions. Visit 1 Enrollment Measurements Week 1 Day 2 the subject will return the 24-hour urine collection and the 24 hour ABPM will be removed. The study medication chlorthalidone will be started. The subject will take study medication for 3 weeks before returning for the next study visit: Visit 2 (Week 3) Day 1 . A three day window will be allowed.

At Visit 2 (Week 3) Day 1 and 2. Biometric measurements: Body Weight and home B/P recordings, start 24 hour Urine collection. Review pill count for compliance, concomitant medications and adverse reactions will be obtained. Day 2: the subject will return the 24-hour urine collection. Review study removal criteria After taking the study medication for three weeks, the subject will return to the CRS unit for Visit 3 End of Study, (Week 7) Day 1 and 2 Visit 3 End of Study, (Week 7) Day 1 and 2. On day 1, Biometric measurements: Body Weight, start 24-h ABPM , Urine studies: start 24 hour Urine collection, safety laboratory evaluations: 8-10AM sitting upright Plasma Aldosterone/Renin Ratio, collect safety labs: bone morphogenetic protein, Mg/phosphorus level, parathyroid hormone, vitamin D level and HbA1c, document pill count, concomitant medications, home blood pressure readings and adverse Reactions. Day 2: the subject will return the 24-hour urine collection and the 24 hour ABPM will be removed If blood pressure is adequately controlled on study medication subject may continue study medication. If blood pressure not adequately controlled on study medication the subject may return to pre-study medication or a medication prescribed by physician.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to participate in study
2. Patients after kidney transplantation> 6 months post-transplant.
3. Age>18 years
4. Home or office Systolic Blood pressure >140 confirmed with daytime 24-h ABPM of average systolic blood pressure >140.
5. Tacrolimus/Cyclosporine therapy with therapeutic trough level based upon historical values
6. Stable renal function for at least 3 months before enrollment.
7. Historical Baseline estimated Glomerular Filtration Rate >30mL/min
8. No more than trace edema on physical examination at time of initial assessment.
9. Receiving optimal doses of ≥ 3 anti-hypertensive medications including furosemide at ≤80mg/d.9.
10. 8-10 in morning sitting Plasma aldosterone Concentration < 15ng/dL and Plasma Renin Activity <0.6ng/mL/h

Exclusion Criteria:

1. Serum sodium<135meq/L based upon historical values
2. Serum potassium<3.5meq/L based upon historical values
3. Poorly controlled diabetes mellitus with HbA1c>9% based upon historical values
4. Already on thiazide
5. Arm circumference >42cm
6. Clinically significant hepatic dysfunction based upon medical history or historical values
7. Two (2) Unsuccessful baseline ABPMs
8. Poor adherence in run-in period as suggested by an unsuccessful 24-h urine collection.
9. DBP≥110 or SBP≥200
10. Allergy to Chlorthalidone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Change from mean baseline systolic blood pressure (by ABPM) between week 0, 1 and 7, ANOVA ABPM at baseline, week 1 and end of the study, Least-squares mean and standard error of the mean for changes in blood pressure measures, | Week 1, week 3, and end of study
  To examine the efficacy of Chlorthalidone as an antihypertensive agent in the treatment of resistant hypertension among stable kidney transplant recipients

OTHER OUTCOMES:
Change in urine studies including urine sodium, chloride and calcium using the non-parametric Wilcoxon test | Week 1, week 3, and end of study
  To examine the efficacy and safety of Chlorthalidone as an antihypertensive agent tin the treatment of resistant hypertension among stable kidney transplant recipients
Adverse events requiring interventions Hypokalemia (K<3meq/L) Hypokalemia (Na<130meq/L r Na<135meq/L accompanied by symptoms, symptomatic Hypotension, rise in serum Creatinine and blood urea nitrogen >2x baseline | Week 1, week 3, and end of study
  To examine the safety of Chlorthalidone as an antihypertensive agent tin the treatment of resistant hypertension among stable kidney transplant recipients

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Gupta, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealtlh University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471